CLINICAL TRIAL: NCT06903208
Title: Radiofrequency Ablation as a Scar-free, Non-operative Approach to Treatment of Superficial Lipomas
Brief Title: RFA for Superficial Lipomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Katherine Fischkoff, Associate Professor of Surgery in Anesthesiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV2254
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lipoma
Keywords: lipoma; ablation; fatty tissue; fatty tumor; scarring; minimally invasive
MeSH Terms: conditions — Lipoma; Cicatrix | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiofrequency ablation (RFA) (Experimental): As this is a single-arm study, all patients enrolled will get the study procedure/treatment of radiofrequency ablation (RFA).
  Interventions: Device: STARMed VIVA Combo RF System

INTERVENTIONS:
Device: STARMed VIVA Combo RF System — RFA is a kind of treatment that uses a long thin needle, called a probe, to melt the lipoma. After numbing the skin with a local anesthetic, using an ultrasound machine as a guide, the study surgeon will insert the probe into the center of the lipoma. The probe will then deliver heat to the lipoma, melting it. The ultrasound is a machine which bounces sound waves to create an image that the study doctor sees on a screen. These ultrasound images will help the study surgeon to accurately guide the probe to the correct location of the lipoma. Once the lipoma is melted, the study surgeon will aspirate any residual liquid out.
  Other Names: Radiofrequency Ablation (RFA)

SUMMARY:
Lipomas are non-cancerous growths of fatty tissue that develop under the skin in approximately 1 in 1000 people, though this number may be higher. While rarely symptomatic, they often cause emotional distress due to the unappealing appearance of the mass. Treatment of unsightly lipomas is excision with local anesthetic in the office or with sedation in the operating room. The recovery period is short and the procedure is low risk; however, the result of the operation is a visible scar over the site of the lipoma. Many patients defer surgical excision because excision of a lipoma is a cosmetic procedure, but the aesthetic outcome is undesirable.

Radiofrequency ablation (RFA) is a technique that applies heat generated by a high frequency, alternating current to soft tissue. The hyperthermia produced by the current causes tissue necrosis that ablates the tissue into which the energy is directed. RFA has been successfully applied to thyroid nodules, pancreatic lesions, esophageal dysplasia and liver tumors. However, the manufacturers of the RFA technology have been focused on its application in pre-malignant and malignant lesions and have not yet considered its application to benign tumors. This study will test the success of RFA for superficial lipomas as a non-surgical option for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Patients with a lipoma <5 cm, above the fascia on the trunk, abdomen or extremities

Exclusion Criteria:

* Lipomas of the face or neck
* Angiolipomas (identified on exam as a firm, mobile, occasionally discolored mass)
* Patients with history of hereditary retinoblastoma, Li-Fraumeni syndrome, familial adenomatous polyposis, neurofibromatosis, tuberous sclerosis and Werner syndrome
* A history of exposure to herbicides, arsenic and dioxin
* A history of radiation treatment for other cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 1 month, 6 months and 12 months post-procedure
  Patient satisfaction will be measured by self-reporting on a Likert scale asking whether they would recommend the procedure: "On a scale of 1 (would not recommend) to 5 (would highly recommend), how likely would you be to recommend RFA treatment of a lipoma to a friend?"
Change in Lesion Volume | Baseline, 1 month, 6 months and 12 months post-procedure
  Lesion volume change from baseline to 1 year.

SECONDARY OUTCOMES:
Complication rate | 1 month, 6 months and 12 months post-procedure
  Number of any complications after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Fischkoff, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States